CLINICAL TRIAL: NCT06183658
Title: Greater-Bay-Area Healthy Aging Brain Study (GHABS): Biomarker- and Neuroimaging-based Study of the Pathophysiology Characterization and Evolutionary Patterns of Alzheimer's Disease
Brief Title: Greater-Bay-Area Healthy Aging Brain Study (GHABS)
Acronym: GHABS
Status: Recruiting | Type: Observational
Sponsor: Shenzhen Bay Laboratory (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Guangdong Basic and Applied Basic Science Foundation (Unknown); Shenzhen Science and Technology Innovation Commission (Unknown)
Responsible Party: Principal Investigator, Tengfei Guo, Principal Investigator, Shenzhen Bay Laboratory
Other Study IDs: YL2023-001
Record Dates: First submitted 2023-11-22; First posted 2023-12-27 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, cerebral spinal fluid, and stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fluids biomarker and neuroimaging of AD diagnosis — Early diagnosis of Alzheimer's disease in South China aging population using fluids biomarker and neuroimaging.

SUMMARY:
The goal of this observational study is to learn about the pathophysiology characterization and evolutionary patterns of Alzheimer's disease (AD) in South China older adults. The primary purposes are as follows:

1. The prevalence and characteristics of AD in South China's aging population
2. Identify novel biomarkers and neuroimaging techniques for early detection and intervention of AD
3. Supporting and fertilizing novel approaches and techniques for early diagnosis and intervention of AD Participants will undergo cognitive assessments, blood sample collection, and genetic testing. Some will undergo CSF collection, stool sample collection, MRI scanning, Aβ PET scanning, and tau PET scanning.

DETAILED DESCRIPTION:
The Greater-Bay-Area Healthy Aging Brain Study (GHABS), a community-based longitudinal cohort study, aimed to characterize of Alzheimer's disease in South China's Aging Population, was launched in May 2021 in Shenzhen. The GHABS project was approved by the Shenzhen Bay Laboratory's and the collaborated hospitals' Ethical Committees. Each participant signed the written informed consent of the GHABS project before enrollment. The participants who met the inclusion and exclusion requirements were informed about the baseline and follow-up examinations. From 2021 to 2026, the GHABS cohort will recruit 1400 individuals aged 55 and older, including 1100 CU older adults, 200 MCI patients, and 100 dementia patients.

All the GHABS participants will undergo cognitive assessments, genetic screening, and blood sample collection. Some will have CSF collection, stool sample collection, MRI scanning, Aβ PET scanning, and tau PET scanning. All baseline examinations will be completed within three months. At follow-up, clinical assessments and blood sample collection will be conducted annually. CSF sample collection, MRI scan, Aβ PET scan, and tau PET scan are evaluated every two years.

ELIGIBILITY:
Inclusion Criteria:

* This project intends to recruit men and women between the ages of 55 and 90. The inclusion criteria are as listed:
* Age 55-90 years old (including 55 and 90 years old). However, people with autosomal dominant and other familial Alzheimer disease (FAD) are not limited by age.
* The score of the Geriatric Depression Scale (GDS) is less than 6 points.
* There is a caregiver who can maintain at least 10 hours of contact per week and can accompany volunteers to the test site for testing.
* Visual and auditory acuity is sufficient for neuropsychological testing. (Including normal corrected vision and hearing)
* Be in good health and are expected to be free of disease interference during the study.
* Volunteers are not pregnant, lactating or have reproductive potential (that is, women must be two years after menopause or undergo sterilization surgery).
* Willingness and ability to participate in longitudinal imaging studies.
* A modified version of the Hachinski Ischemic scores less than or equal to 4.
* Have completed grade 6 education or have good work experience (sufficient to rule out mental retardation).
* Must be able to speak Mandarin fluently.
* Willing to undergo multiple 3T MRI scans and at least two PET scans.
* Agree to collect blood for genomic analysis (including GWAS sequencing and other analyses), AD risk and protective genes such as apolipoprotein E (APOE), klotho, etc., and biological sample storage.
* Agree to collect blood for biomarker detection.
* Agree to share genomic data and biomarker samples.

Exclusion Criteria:

* MRI brain scan screening reveals infection, infarction or other focal lesions or multiple lacunes or lacunes in key memory structures.
* Any volunteers who do not meet the MRI scan requirements, including having a cardiac pacemaker, eyes, skin or metal fragments or foreign bodies in the body.
* Severe depression, bipolar affective disorder described in DSM-IV in the past year.
* Psychotic features, agitation or behavioral problems that may lead to difficulty complying with the protocol content in the past 3 months.
* Currently using medication to treat obsessive-compulsive disorder or attention deficit disorder.
* History of schizophrenia (meeting DSM-IV criteria).
* History of alcohol or drug abuse or dependence within the past 2 years (metting DSM-IV criteria).
* Any major systemic disease or unstable physical condition that may make longitudinal research difficult.
* Clinically significant abnormalities of B12 or TFTs may interfere with the study, low B12 will be excluded.
* Currently using certain psychoactive medications (e.g., certain antidepressants, neuro-depressants, chronic anxiolytics, or sedative-hypnotics). Currently using warfarin or other anticoagulants such as dabigatran, rivaroxaban, and apixaban (except lumbar puncture).
* Use of prohibited drugs.
* Simultaneously participating in other clinical studies involving neuropsychiatry.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The GHABS cohort will recruit 1400 individuals aged 55 and older, including cognitively unimpaired older adults, subjective cognitive decline, mild cognitive impairment, and dementia.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Longitudinal changes of cognitive function _ ADAS-Cog | An average of 1 year
  Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog)
Longitudinal changes of cognitive function _ MMSE, the Chinese version | An average of 1 year
  Mini-mental State Examination (MMSE, the Chinese version)
Longitudinal changes of cognitive function _ MoCA-Basic | An average of 1 year
  Montreal Cognitive Assessment Basic (MoCA-Basic)
Longitudinal functional and behavioral function _ CDR | An average of 1 year
  Clinical Dementia Rating (CDR)
Longitudinal functional and behavioral function _ NPI | An average of 1 year
  Neuropsychiatric Inventory (NPI)
Longitudinal functional and behavioral function _ GDS | An average of 1 year
  Geriatric Depression Scale (GDS)
Longitudinal functional and behavioral function _ FAQ | An average of 1 year
  Function Activities Questionnaire (FAQ)
Longitudinal functional and behavioral function _ ADL | An average of 1 year
  Activity of Daily Living Scale (ADL)
Longitudinal functional and behavioral function _ PSQI | An average of 1 year
  Pittsburgh sleep quality index (PSQI)
Longitudinal functional and behavioral function _ RBDSQ | An average of 1 year
  REM sleep behavior disorder screening questionnaire (RBDSQ)

SECONDARY OUTCOMES:
Longitudinal changes of plasma biomarkers | An average of 1 year
  Longitudinal changes of disease status as categorized by plasma biomarkers of Alzheimer's diseases over time.
Longitudinal changes of CSF biomarkers | An average of 2 years
  Longitudinal changes of disease status as categorized by CSF biomarkers of Alzheimer's diseases over time.
Longitudinal changes in neuroimaging _ MRI images | An average of 2 years
  Longitudinal change in brain structure using magnetic resonance imaging (MRI)
Longitudinal changes in neuroimaging _ amyloid PET images | An average of 2 years
  Longitudinal changes in amyloid deposition
Longitudinal changes in neuroimaging _ tau PET images | An average of 2 years
  Longitudinal changes in tau deposition

OTHER OUTCOMES:
Correlation of microbiome to Alzheimer's Disease | 1 time sampling
  Correlation of microbiome to Alzheimer's Disease via relative abundance found in gut microbiome study. These data will then be correlated to Alzheimer's disease state

CONTACTS AND LOCATIONS:
Overall Officials: Tengfei Guo, Ph.D., Principal Investigator — Shenzhen Bay Laboratory
Locations (1):
- Shenzhen Bay Laboratory, Shenzhen, Other, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT06183658/ICF_000.pdf